CLINICAL TRIAL: NCT03603717
Title: Improving Sleep as a Strategy to Reduce Suicide Risk Among At-Risk Veterans: A Real World Clinical Trial
Brief Title: RCT of Brief CBT-I in Primary Care Veterans With Suicidal Thoughts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IIR 16-055; I01HX002183-01A2 (NIH)
Record Dates: First submitted 2018-07-19; First posted 2018-07-27 (Actual); Results first posted 2024-06-17 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2023-12

CONDITIONS: Insomnia; Suicidal Ideation
Keywords: insomnia; suicidal ideation; depression; posttraumatic stress disorder; cognitive behavioral therapy for insomnia; sleep; suicide
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Suicidal Ideation; Depression; Stress Disorders, Post-Traumatic; Suicide | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Two parallel study arms: (1) cognitive behavioral therapy for insomnia (the experimental condition) and (2) sleep hygiene (the control condition).
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be informed that they are receiving one of two non-medication sleep interventions. Assessors are blinded to study condition. Study staff entering data will be blinded to condition. It is not possible to blind staff delivering the interventions. The PI's are providing some supervision of the interventionists, so they will be unblinded for those participants they supervise interventionists on.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CBT-I (Experimental): Four individual sessions that will last approximately 15-30 minutes each across a 6-week time period, with the option to deliver sessions over the telephone as necessary.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia
- Sleep Hygiene (Active Comparator): Four individual sessions that will last 15-30 minutes each across a 6-week time period, with the option to deliver sessions over the telephone as necessary.
  Interventions: Behavioral: Sleep Hygiene

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia — The intervention will consist of a standard, structured, multi-component intervention for insomnia that includes sleep education, sleep hygiene, sleep restriction, stimulus control, and cognitive therapy.
  Arms: CBT-I
Behavioral: Sleep Hygiene — The intervention will include basic psychoeducation about sleep, discussion of sleep hygiene factors that disrupt and improve sleep, setting sleep hygiene goals, and developing action steps to achieve those goals.
  Arms: Sleep Hygiene

SUMMARY:
There is a strong association between insomnia and suicidal thoughts and behaviors. Insomnia also frequently co-occurs with other common conditions associated with suicide such as depression and posttraumatic stress disorder. This project focuses on improving sleep as a novel suicide prevention strategy that can be delivered to a broad range of Veterans. The study will examine how Cognitive Behavioral Therapy for Insomnia, an efficacious treatment for insomnia, may reduce suicidal thoughts in Veterans who also suffer from co-occurring conditions when delivered by integrated primary care clinicians.

DETAILED DESCRIPTION:
Anticipated Benefit to VA Healthcare The proposed study will establish the feasibility and effectiveness of treating insomnia in the primary care environment as a suicide prevention strategy. By treating insomnia, a common problem that is both a risk factor for suicide and highly prevalent in common conditions associated with suicide such as depression and posttraumatic stress disorder (PTSD), the investigators expect to reduce the severity of suicidal ideation (SI) among Veterans experiencing SI, insomnia and a co-occurring condition.

Project Background Suicide is the tenth leading cause of death in the U.S., is a major concern of the Department of Veterans Affairs (VA) and occurs at elevated rates among Veterans. Veterans with common chronic conditions such as PTSD and depression are at increased risk for suicide. Although evidence-based treatments exist for these conditions, a significant number of Veterans do not engage in or complete such treatments leaving them at higher risk for suicide.

This application builds upon VA funded pilot work that demonstrated the feasibility of delivering a brief version of cognitive-behavioral therapy for insomnia (CBT-I) within primary care to Veterans experiencing SI. The pilot data suggest that the investigators' brief, primary-care based insomnia treatment was delivered with high fidelity, acceptable to Veterans and associated with significant reductions in insomnia and depression symptoms, and reduced SI intensity. The next stage of this program of research is to establish the feasibility of delivering the brief, primary care based, insomnia intervention utilizing primary care-mental health integration (PC-MHI) clinicians (as opposed to research staff) and to establish the effectiveness of the intervention on reducing the severity of factors that contribute to suicide risk and to improve other clinical markers in a definitive trial.

Project Objectives The ultimate goal of the broader program of research is to reduce suicide among Veterans by intervening upon sleep disturbance as a modifiable risk factor for suicide. In this application the investigators focus on insomnia, which is the most common sleep disorder among Veterans and is robustly associated with suicidal thoughts and behaviors.

The primary objective of this proposed clinical trial is to test whether (and how) using brief behavioral insomnia treatment can not only improve sleep, but reduce other risk factors for suicide including the severity of depression, PTSD and suicidal ideation among Veterans at risk for suicide. Secondary objectives are to: (1) gather initial data on barriers and facilitators to implementation to aid future implementation efforts in VA primary care and (2) determine if the intervention improves attitudes towards psychotherapy treatments that address the co-morbid conditions.

Project Methods In order to achieve these objectives the investigators will conduct a real-world, randomized clinical trial among 240 Veterans experiencing either co-occurring depression or PTSD recruited from primary clinics at three VA sites. These Veterans, who will also endorse SI and insomnia, will be randomized to receive either a brief course of CBT-I or a sleep hygiene intervention of similar length. Assessments of suicidal thoughts and behaviors, insomnia, depression, and PTSD will be conducted at baseline, post-treatment, and every 6 weeks thereafter until 6 months post-treatment. Mixed effects modeling and structured equation modeling will be applied to determine how improvements in sleep and other symptoms (e.g. depression, PTSD) contribute to reductions in SI severity. In addition, the investigators will collect, code and analyze participant and provider feedback to assess barriers and facilitators of implementation in real-world clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Veteran seeking or receiving services at the Canandaigua, Buffalo or Syracuse VA Medical Centers
* Demonstrate understanding of informed consent
* Endorse current death/suicidal ideation on item 9 of the Patient Health Questionnaire-9
* An Insomnia Severity Index score > 10 with trouble sleeping 3 months and at least 1 insomnia-related daytime consequence
* Either:

  * [a] a current diagnosis of Major Depressive Disorder, Depression not otherwise specified or PTSD
  * [b] a score of > 16 on the Patient Health Questionnaire for Depression (PHQ-9) or a score > 46 on the PTSD Symptom Checklist
* If using psychotropic medications the dosage must be stable

Exclusion Criteria:

* History of serious mental illness such as schizophrenia, Bipolar I or II disorder, or current psychiatric conditions such as psychosis, mania, dementia or cognitive impairment
* A suicide attempt within the last 6 months or [report of SI with active plan or intent in the past month]
* Currently engaged in inpatient or partial hospitalization programs
* Recent substance dependence disorder with < 6 months abstinence
* Narcolepsy
* Circadian rhythm disorders
* Restless legs syndrome
* Untreated sleep apnea based upon chart review
* A sleep disorders screening questionnaire and the STOP-BANG sleep apnea questionnaire

  * Sleep medications are not exclusionary, but participants using them must still meet insomnia criteria

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 283 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wilfred R. Pigeon, PhD, Principal Investigator — VA Finger Lakes Healthcare System, Canandaigua, NY
Locations (3):
- United States (3):
  - VA Western New York Healthcare System, Buffalo, NY, Buffalo, New York
  - VA Finger Lakes Healthcare System, Canandaigua, NY, Canandaigua, New York
  - Syracuse VA Medical Center, Syracuse, NY, Syracuse, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited by a letter from their primary care physician from three Department of Veterans Affairs Medical Centers and then screened by telephone by study staff between January 2019 and November 2022. The first participant was enrolled on February 8, 2019 and the last participant enrolled in November 2022.
Pre-assignment Details: A total of 283 participants were enrolled in the study and completed the baseline assessment. Of these, 83 did not meet eligibility criteria and 6 eligible participants withdrew prior to randomization. As a result, 194 participants were randomized.
Period: Overall Study
Arm/Group | CBT-I | Sleep Hygiene
Started | 98 | 96
Completed | 62 | 66
Not Completed | 36 | 30
Not completed — Lost to Follow-up | 20 | 20
Not completed — Withdrawal by Subject | 16 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CBT-I | Sleep Hygiene | Total
Number analyzed (Participants) | 98 | 96 | 194
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.49 (14.50) | 51.51 (12.83) | 51.50 (13.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 24 | 45
  Male | 77 | 72 | 149
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 12 | 18
  Not Hispanic or Latino | 91 | 84 | 175
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 3
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 9 | 14
  White | 81 | 79 | 160
  More than one race | 7 | 8 | 15
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 98 | 96 | 194
Insomnia Severity Index Change [Mean (Standard Deviation); unit: units on a scale] — Rated on a 0-4-point scale with a total score range of 0-28 where higher scores indicate greater severity
  units on a scale | 19.52 (4.14) | 18.58 (4.10) | 19.06 (4.14)
Scale for Suicidal Ideation Change [Mean (Standard Deviation); unit: units on a scale] — Rated on a 0-2 point scale with a total score range of 0-38 where higher scores indicate greater severity
  units on a scale | 3.21 (4.73) | 3.88 (5.86) | 3.54 (5.32)
PTSD Symptom Checklist-DSM 5 Change [Mean (Standard Deviation); unit: units on a scale] — Rated on a 0-4 point scale with a total score range of 0-80 where higher scores indicate greater severity
  units on a scale | 45.29 (13.48) | 41.53 (14.97) | 43.43 (14.32)
Patient Health Questionnaire-Depression Change [Mean (Standard Deviation); unit: units on a scale] — Rated on a 0-3 point scale with a total score range of 0-27 where higher scores indicate greater severity
  units on a scale | 15.88 (4.93) | 14.47 (5.24) | 15.18 (5.12)

OUTCOME MEASURES:

1. Primary Outcome: Insomnia Severity Index Change
Description: The Insomnia Severity Index (ISI) is a 7-item self-report measure of insomnia symptoms. Each item is rated on a 0-4-point scale with a total score range of 0-28 where higher scores indicate greater severity.
Time Frame: Baseline (Week 0) and 6 Month follow-up (Week 30)
Population: All participants who were assigned to the arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT-I | Sleep Hygiene
Number analyzed (Participants) | 98 | 96
score on a scale | 8.54 (6.03) | 11.88 (6.36)
Statistical Analysis 1: Comparison: CBT-I vs Sleep Hygiene; Test type: Superiority; p < 0.01, Mixed Models Analysis

2. Secondary Outcome: Scale for Suicidal Ideation Change
Description: The Scale for Suicidal Ideation is a clinician administered scale with 19-items related to suicidal ideation. Each item is rated on a 0-2 point scale with a total score range of 0-38 where higher scores indicate greater severity.
Time Frame: Baseline (Week 0) and 6 Month follow-up (Week 30)
Population: All participants who were assigned to study arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT-I | Sleep Hygiene
Number analyzed (Participants) | 98 | 96
score on a scale | 1.08 (2.08) | 3.10 (5.12)
Statistical Analysis 1: Comparison: CBT-I vs Sleep Hygiene; Test type: Superiority; p = 0.03, Mixed Models Analysis

3. Secondary Outcome: PTSD Symptom Checklist-DSM 5 Change
Description: The PTSD Symptom Checklist-DSM 5 version is a 20-item self-report measure of PTSD symptoms. Each item is rated on a 0-4 point scale with a total score range of 0-80 where higher scores indicate greater severity.
Time Frame: Baseline (Week 0) and 6 Month follow-up (Week 30)
Population: All participants who were assigned to study arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT-I | Sleep Hygiene
Number analyzed (Participants) | 98 | 96
score on a scale | 29.68 (18.02) | 29.94 (17.62)
Statistical Analysis 1: Comparison: CBT-I vs Sleep Hygiene; Test type: Superiority; p = 0.84, Mixed Models Analysis

4. Secondary Outcome: Patient Health Questionnaire-Depression Change
Description: The Patient Health Questionnaire-Depression is a 9-item self-report measure of depression symptoms. Each item is rated on a 0-3 point scale with a total score range of 0-27 where higher scores indicate greater severity.
Time Frame: Baseline (Week 0) and 6 Month follow-up (Week 30)
Population: All participants who were assigned to study arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT-I | Sleep Hygiene
Number analyzed (Participants) | 98 | 96
score on a scale | 8.92 (6.03) | 11.33 (6.48)
Statistical Analysis 1: Comparison: CBT-I vs Sleep Hygiene; Test type: Superiority; p = 0.01, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 30 weeks
Arm/Group | CBT-I | Sleep Hygiene
All-Cause Mortality (participants affected / at risk) | 0/98 | 0/96
Serious Adverse Events (participants affected / at risk) | 3/98 | 4/96
Other Adverse Events (participants affected / at risk) | 2/98 | 0/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CBT-I (N=98) | Sleep Hygiene (N=96)
Hospitalization (Cardiac disorders) | 1 (1) | 2 (2)
Hospitalization (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hospitalization (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hospitalization (Psychiatric disorders) | 1 (1) | 0 (0) — Suicide attempt (overdose)
hospitalization (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CBT-I (N=98) | Sleep Hygiene (N=96)
Emergency room visit for migraine headache (Nervous system disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-18): https://cdn.clinicaltrials.gov/large-docs/17/NCT03603717/Prot_SAP_000.pdf